CLINICAL TRIAL: NCT04825145
Title: Preeclampsia and Contact Activation
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Collaborators: Region of Southern Denmark (Other); OPEN (Unknown); Lida og Oskar Nielsens Fond (Unknown); Esbjerg Fonden (Other); Gangsted Fonden (Unknown)
Responsible Party: Principal Investigator, Anne Cathrine Meldgaard Godtfredsen, Principal investigator, medical doctor, phd student, University of Southern Denmark
Other Study IDs: s-20190142
Record Dates: First submitted 2021-03-25; First posted 2021-04-01 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Preeclampsia; CAS; Misfolding Disease, Protein
Keywords: Contact activation system, PAI-2
MeSH Terms: conditions — Pre-Eclampsia; Proteostasis Deficiencies | interventions — Pregnancy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Preeclamptic women: Pregnant women who is diagnosed with preeclampsia during anytime of pregnancy.
  Interventions: Other: Pregnancy
- Healthy pregnant women: Pregnant women without preeclampsia. Will be matched for body mass index, gestational age and age.

INTERVENTIONS:
Other: Pregnancy — Pregnancies complicated by preeclampsia
  Groups: Preeclamptic women

SUMMARY:
Preeclampsia (PE) affects approximately 5% of all pregnancies with 2,500 cases registered annually in Denmark. PE is characterized by incomplete modelling of the spiral arteries of the uterus, hypertension, inflammation, hypercoagulability and proteinuria. Neonatal complications and increased cardiovascular risk are common features of the syndrome.

PE shares pathophysiologic features with recognized protein misfolding disorders and misfolded proteins are present in urine from women with PE. Misfolded proteins are potent activators of the contact system (CAS) which is involved in inflammation, coagulation and fibrinolysis.

Plasminogen activator inhibitor 2 (PAI-2) regulates important fibrinolytic processes in the placenta. The oxidative milieu characterizing PE may trigger misfolding of PAI-2 which then loose inhibitory capacity, but gain CAS-activating capacity. Thus, misfolding of PAI-2 may affect the fibrinolytic system in the placenta and compromise the modelling of the spiral arteries. Moreover, misfolded PAI-2 may contribute to the hypercoagulability and the inflammatory conditions characterizing women with PE.

The aim of the present study is i) to characterize CAS in women with PE, ii) to study the CAS-activating capacity of misfolded PAI-2 and iii) to develop and apply immunochemical methods for determination of native and misfolded PAI-2 in plasma.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women developing preeclampsia

Exclusion Criteria:

* Healthy pregnant women

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Preeclamptic women anytime of pregnancy compared to healthy pregnant women (control) at the same gestational age, with matching BMI and age.
Sampling Method: Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
The Contact Activation System (CAS) | 3 years
  Biomarkers for the CAS in plasma Coagulation factor XII antigen/activity, High molecular weight kininogen (HK), Truncated (HK), Prekallikrein antigen, kallikrein generation, C1-esterase inhibitor, alpha-2-macroglobulin, Fast form alpha-2-macroglobulin, Thrombin generation,
Misfolded Plasminogen activator inhibitor 2 (PAI-2) | 3 years
  Biomarkers for misfolded PAI-2 in plasma Native PAI-2 antigen, Misfolded PAI-2, Native PAI-1 antigen,

CONTACTS AND LOCATIONS:
Overall Officials: Jørgen B Gram, Professor, Study Director — University of Southern Denmark
Locations (1):
- The Unit for Thrombosis Research, University of Southern Denmark, Esbjerg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Godtfredsen AC, Palarasah Y, Dolleris BB, Jorgensen JS, Sidelmann JJ, Gram JB. Increased contact activated endogenous thrombin potential in pregnant women with preeclampsia. Blood Coagul Fibrinolysis. 2024 Jan 1;35(1):1-7. doi: 10.1097/MBC.0000000000001269. Epub 2023 Nov 30. PMID 38051647

DOCUMENTS (1):
  • Study Protocol (2020-01-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT04825145/Prot_000.pdf